CLINICAL TRIAL: NCT00446082
Title: A Phase I, Multicenter, Open-label, Randomized Study Assessing the Pharmacokinetics, Safety, and Tolerability of Monthly Doses of Pasireotide i.m. LAR Injection in Patients With Acromegaly and Patients With Carcinoid Disease
Brief Title: Study of Pasireotide Long Acting Release (LAR) Injection in Patients With Acromegaly and Patients With Carcinoid Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230C2110; 2005-003348-75 (EudraCT Number)
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-11

CONDITIONS: Carcinoid Tumor; Acromegaly
Keywords: Refractory/ resistant carcinoid disease; acromegaly; adults; pasireotide LAR; somatostatin analogue; SOM230; pharmacokinetics; Refractory or resistant carcinoid disease and acromegaly
MeSH Terms: conditions — Carcinoid Tumor; Acromegaly | interventions — pasireotide

ARMS (1):
- SOM230 LAR (Experimental)
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide

SUMMARY:
This study will assess the pharmacokinetic profile and the safety/tolerability profile of single and monthly doses of pasireotide LAR intramuscular (i.m.) injection in patients with acromegaly and patients with carcinoid disease

ELIGIBILITY:
Inclusion criteria for patients with acromegaly:

* Male or female patients between 18 and 80 years
* Patients with acromegaly due to a pituitary adenoma with elevated GH and IGF-1 concentrations

Exclusion criteria for patients with acromegaly:

* Patients with compression of the optic chiasm causing any visual field defect
* Specific criteria apply for patients who have received certain types of therapies such as radiotherapies, surgeries, chemo- or immunotherapies in the months prior to study start
* Female patients who are pregnant or lactating

Inclusion criteria for patients with carcinoid disease:

* Male or female patients aged ≥18 years
* Patients with histologically confirmed, metastatic carcinoid tumors of the digestive system
* Patients with elevation of chromogranin-A (CgA) and/or serotonin
* Patients who are not adequately controlled by somatostatin analogues

Exclusion criteria for patients with carcinoid disease:

* Specific criteria apply for patients who have received certain types of therapies such as radiotherapies, surgeries, chemo- or immunotherapies in the months prior to study start
* Female patients who are pregnant or lactating

Other protocol-defined in- and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Determination of the pharmacokinetic profile of single and monthly doses of pasireotide LAR i.m. injection | Baseline, D7, D35, D63
  in patients with acromegaly and in patients with carcinoid disease

SECONDARY OUTCOMES:
To explore the pharmacodynamic profile of single and monthly doses of pasireotide LAR i.m. injection | Baseline, D7, D35, D63
  in patients with acromegaly and in patients with carcinoid disease.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Chair — Novartis
Locations (16):
- United States (4):
  - Cedars Sinai Medical Center SC - 4, Los Angeles, California
  - Stanford University Medical Center Stanford Cancer Center (3), Stanford, California
  - H. Lee Moffitt Cancer Center & Research Institute Dept.of H.LeeMoffittCC&RI(1), Tampa, Florida
  - University of Texas/MD Anderson Cancer Center Gastrointestinal Med. Oncology, Houston, Texas
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Canada (3):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Oslo, Norway

REFERENCES:
- [Result] Petersenn S, Bollerslev J, Arafat AM, Schopohl J, Serri O, Katznelson L, Lasher J, Hughes G, Hu K, Shen G, Resendiz KH, Giannone V, Beckers A. Pharmacokinetics, pharmacodynamics, and safety of pasireotide LAR in patients with acromegaly: a randomized, multicenter, open-label, phase I study. J Clin Pharmacol. 2014 Nov;54(11):1308-17. doi: 10.1002/jcph.326. Epub 2014 May 24. PMID 24800725
- See also: Novartis Clinical Trial Results for CSOM230C2110 — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12987